CLINICAL TRIAL: NCT02448355
Title: Ocular Effects of Carotid Endarterectomy A Cohort Longitudinal Study
Brief Title: Ocular Effects of Carotid Endarterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, joel hanhart, MD, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: hanhart1
Record Dates: First submitted 2014-11-28; First posted 2015-05-19 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Choroid; Carotid Stenosis; Carotid Endarterectomy
Keywords: OCT
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient undergoing carotid endarterectomy (Experimental): All patients undergoing carotid endarterectomy in Shaare Zedek Medical Center Visual acuity measurement (Snellen) SS-OCT (DRI-Atlantis, Topcon) 3-dimensional scanning protocol with 3 μm axial resolution and a speed of 100,000 A-scans per second. 256 B-scans to be taken on an area of 12 × 9 μm.
  * On pre-op visit (Monday)
  * Day 1 post-surgery
  * Discharge day
  * Week 1 post-surgery
  * Month 1 post-surgery
  Interventions: Device: OCT swept source DRI-Atlantis, Topcon

INTERVENTIONS:
Device: OCT swept source DRI-Atlantis, Topcon — 3-dimensional scanning protocol with 3 μm axial resolution and a speed of 100,000 A-scans per second. 256 B-scans to be taken on an area of 12 × 9 μm.

SUMMARY:
All patients undergoing carotid endarterectomy in Shaare Zedek Medical Hospital, during about 1 year, will be offered to participate.

Retinal and choroidal structural changes will be assessed using swept-source OCT technology

ELIGIBILITY:
Inclusion Criteria:

* Carotid stenosis requiring surgical management

Exclusion Criteria:

* Ocular conditions: media opacities precluding fundus visualization, bilateral no-light perception
* Ocular surgery within 6 months prior to endarterectomy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in choroidal thickness | one year
  Change in choroidal thickness (microns) on OCT pictures

SECONDARY OUTCOMES:
Visual acuity | One year
  Visual acuity as assessed by Snellen chart
Retinal changes | One year
  Analysis of OCT pictures